CLINICAL TRIAL: NCT02440451
Title: Improving Facial Expression Identification in ASD: a Real-time fMRI Neurofeedback Approach
Brief Title: Rt-fMRI NF Intervention Study in ASD
Acronym: NF-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, MD, PhD, University of Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBILI-VB-2015-02
Record Dates: First submitted 2015-04-24; First posted 2015-05-12 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurofeedback using BCI (Experimental): 16 (13 + 3 in case of dropoffs) ASD subjects
  Interventions: Device: Neurofeedback using BCI

INTERVENTIONS:
Device: Neurofeedback using BCI — This group will undergo five sessions of neurofeedback intervention in the fMRI scanner. Each subject will also undergo neuropsychological evaluations before the first neurofeedback session (week 0) and after the last neurofeedback session (week 7). The first four sessions are weekly while the last one is one month later. The intervention will take a total of four months. Follow up will be performed in the the first week and 6 months after the last intervention session.

SUMMARY:
This study aims to demonstrate that fMRI neurofeedback training improves the identification and comprehension of emotional facial expressions (and overall social behaviour) in subjects with ASD.

The intervention setup provides structured presentation of emotional facial expressions and the associated tools for mental imagery. The investigators hypothesize that the accomplishment of the proposed competence training improves the subjects ability to comprehend facial expressions, identify emotions and be able to correctly express them.

Intervention Type is a Device (brain computer interface using brain imaging signals) and the specific Intervention Name is Neurofeedback.

Structure: (1) initial eligibility screening, (2) pre-intervention (first week of study, baseline outcome measures and additional evaluations), (3) intervention process (8 weeks), (4) post-intervention (outcome measures and additional evaluations), and (5) follow-up (outcome measures at 6 months).

DETAILED DESCRIPTION:
Clinical research has demonstrated that ASD children have deficits in the identification and interpretation of the emotional and mental state of others (Baron-Cohen 2001). An important skill to this end (impaired in ASD patients), is to appropriately recognize and discriminate emotional expressions.

The main brain regions involved in face processing the inferior occipital gyri, lateral portion of the fusiform gyrus (especially a region deemed the fusiform face area or FFA), and posterior superior temporal sulcus (pSTS) (Haxby et al. 2000). STS plays a key role on several basic aspects in social information processing, and deficits in ASD have been found associated to this region.

The purpose of the study is to determine the effect of neurofeedback considering a social cognition brain region (i.e. pSTS) on the identification of facial expressions in ASD patients. The intervention comprehends seven BCI sessions spread over four months. The first four sessions are weekly, and the rest monthly. In each session, the subjects are asked to imagine different facial expressions and their brain activity (i.e. BOLD activation in the pSTS region) is interpreted and used to estimate a feedback signal.The hypothesis is that the training induced up-regulation of the target region, improves clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnostic results for ASD in:

Autism Diagnostic Interview-Revised; Autism Diagnostic Observation Schedule; The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.

Exclusion Criteria:

* Global Intelligence Quotient < 80
* Associated medical condition such as epilepsy, neurocutaneous or other genetic syndromes, or other usual comorbidity in ASD samples

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel S Castelo-Branco, M. D., PhD., Principal Investigator — IBILI - Institute for Biomedical Imaging in Life Sciences

REFERENCES:
- [Background] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Background] Haxby JV, Hoffman EA, Gobbini MI. The distributed human neural system for face perception. Trends Cogn Sci. 2000 Jun;4(6):223-233. doi: 10.1016/s1364-6613(00)01482-0. PMID 10827445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants, mainly recruited on a collaborative effort between the Pediatrics Hospital of Coimbra and local ASD associations, were invited for an fMRI neurofeedback feasibility clinical trial study in ASD. All participants had normal or corrected to normal vision. ). The first participant was recruited in February 2016.
Pre-assignment Details: There was no significant events after participant enrollment, before group assignment.
Groups:
- Neurofeedback Using BCI: 16 (13 + 3 in case of dropoffs) ASD subjects
  Neurofeedback (BCI using neuroimaging): This group will undergo five sessions of neurofeedback intervention in the fMRI scanner. Each subject will also undergo neuropsychological evaluations before the first neurofeedback session (week 0) and after the last neurofeedback session (week 7). The first four sessions are weekly while the last one is one month later. The intervention will take a total of four months. Follow up will be performed in the the first week and 6 months after the last intervention session.
Period: Overall Study
Arm/Group | Neurofeedback Using BCI
Started (Started the intervention protocol.) | 15
Completed (Completed the intervention protocol.) | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The number of participants is similar to the assigned in the participant flow.
Arm/Group | Neurofeedback Using BCI
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 19.92 [16.83 to 29.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Portugal | 15
FEEST - Facial Expression of Emotion: Stimuli and Tests [Mean (Standard Deviation); unit: units on a scale] — The Emotion Hexagon Test from Facial expressions of emotion: Stimuli and Test (FEEST) represents the primary outcome measure. The test uses 30 computer-manipulated images of faces from the Ekman and Friesen series to test recognition of basic emotions - anger, disgust, fear, happiness, sadness and surprise.Here we report the total score. The results are converted to a score of min.0 and max.120 correct for recognition of all six emotions. The higher the score, better is the ability to recognize emotions.
  units on a scale | 98 (19.30)
ATEC - Autism Treatment Evaluation Checklist [Mean (Standard Deviation); unit: units on a scale] — Autism Treatment Evaluation Checklist (ATEC) evaluates the effectiveness of autism treatments - a 1-page form designed to be completed by parents or caretakers. It consists of 4 subtests: I. Speech/Language Communication (14 items, min.0-max.28); II. Sociability (20 items, min.0-max.40); III. Sensory/Cognitive Awareness (18 items, min.0-max.36); and IV. Health/Phys./Behavior (25 items, min.0-max.75). Total score (sum) ranges from min.0-max.179.
  The results reported here correspond to the total ATEC score to be used for comparison at a later date. The lower the score, the fewer the problems.
  units on a scale | 36.6 (13.94)
VABS - Vineland Adaptive Behaviour Scale [Mean (Standard Deviation); unit: units on a scale] — The Vineland Adaptive Behaviour Scale (VABS) is a semi-structured interview designed to assess global adaptive functioning, composed by 3 main domains: Communication COM, Daily Living Skills DLS and Socialization SOC (all reported here in terms of standard scores as described in the VABS manual, i.e. mean 100 and standard deviation 15).
  The Adaptive Behaviour Composite ABC (total score, also reported here) is the sum of the raw scores from the three main domains. These are transformed in standard scores (m.=100;std.=15).
  The higher the score, better is the adaptive behavior.
  units on a scale
    Baseline [VABS COM] | 70.6 (15.65)
    Baseline [VABS DLS] | 74 (17.15)
    Baseline [VABS SOC] | 63.4 (14.21)
    Baseline [VABS ABC] | 63.4 (13.52)

OUTCOME MEASURES:

1. Primary Outcome: FEEST - Facial Expression of Emotion: Stimuli and Tests
Description: The Emotion Hexagon test represents the primary outcome measure. The assessment based on this test will be performed before (baseline), after the intervention - endpoint 1 (at 8 weeks) and at the 6 months follow-up. The Emotion Hexagon test uses stimuli of graded difficulty, created using computer image manipulation techniques (morphing is used to modify photographs from the Ekman and Friesen (1976) series, creating examples that lie close to or more distant from the prototype expression). The 120 test trials with unambiguous stimuli (4 pictures for each of the 6 emotions across the 5 test blocks) can be used to derive an overall (total) score out of a possible maximum of 120 expressions correctly recognized.
Time Frame: 8 weeks (Endpoint 1) plus 6 months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurofeedback Using BCI
Number analyzed (Participants) | 15
units on a scale
  Endpoint 1 | 100.27 (19.29)
  6 months follow-up | 100.79 (20.01)

2. Secondary Outcome: ATEC - Autism Treatment Evaluation Checklist
Description: Autism Treatment Evaluation Checklist (ATEC) evaluates the effectiveness of autism treatments - a 1-page form designed to be completed by parents or caretakers. It consists of 4 subtests: I. Speech/Language Communication (14 items, min.0-max.28); II. Sociability (20 items, min.0-max.40); III. Sensory/Cognitive Awareness (18 items, min.0-max.36); and IV. Health/Phys./Behavior (25 items, min.0-max.75). Total score (sum) ranges from min.0-max.179.
  The results reported here correspond to the total ATEC score to be used for comparison at a later date. The lower the score, the fewer the problems.
Time Frame: 8 weeks (Endpoint 1) plus 6 months follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurofeedback Using BCI
Number analyzed (Participants) | 15
units on a scale
  Endpoint 1 | 32 (14.66)
  6 months follow-up | 19.64 (8.13)

3. Secondary Outcome: VABS - Vineland Adaptive Behaviour Scale
Description: The Vineland Adaptive Behaviour Scale (VABS) is a semi-structured interview designed to assess global adaptive functioning, composed by 3 main domains: Communication COM, Daily Living Skills DLS and Socialization SOC (all reported here in terms of standard scores as described in the VABS manual, i.e. mean 100 and standard deviation 15).
  The Adaptive Behaviour Composite ABC (total score, also reported here) is the sum of the raw scores from the three main domains. These are transformed in standard scores (m.=100;std.=15).
  The higher the score, better is the adaptive behavior.
Time Frame: 8 weeks (Endpoint 1) plus 6 months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurofeedback Using BCI
Number analyzed (Participants) | 15
units on a scale
  Endpoint 1 [VABS COM] | 74.87 (14.95)
  Endpoint 1 [VABS DLS] | 76.93 (16.46)
  Endpoint 1 [VABS SOC] | 66.73 (16.42)
  Endpoint 1 [VABS ABC] | 67.13 (15.22)
  6 months follow-up [VABS COM] | 79.79 (13.69)
  6 months follow-up [VABS DLS] | 83.14 (17.00)
  6 months follow-up [VABS SOC] | 71.43 (15.36)
  6 months follow-up [VABS ABC] | 73.57 (13.67)

4. Other Pre Specified Outcome: POMS - Profile of Mood States
Time Frame: 8 weeks (Endpoint 1) plus 6 months follow-up
Reporting Status: Not Posted

5. Other Pre Specified Outcome: HADS - Hospital Anxiety & Depression Scale
Description: 24-item scale (7 depression & 7 anxiety items)
Time Frame: 8 weeks (Endpoint 1) plus 6 months follow-up
Reporting Status: Not Posted

6. Other Pre Specified Outcome: BDI - Beck Depression Inventory
Description: 21-item measure of clinical depression
Time Frame: 8 weeks (Endpoint 1) plus 6 months follow-up
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Debriefing Interview Questionnaire
Description: Covers: strategies; general experience of the process; adverse effects;
Time Frame: 8 weeks (Endpoint 1)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months (from baseline until 6 months follow-up assessment)
Arm/Group | Neurofeedback Using BCI
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT02440451/SAP_000.pdf
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT02440451/Prot_001.pdf